CLINICAL TRIAL: NCT00428571
Title: Laparoscopic Bariatric Surgery for Treatment of Type 2 Diabetes in Obese Patients With End Organ Damage: A Prospective Randomized Controlled Pilot Study
Brief Title: Laparoscopic Bariatric Surgery to Treat Type 2 Diabetes in Obese Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Mehran Anvari, Dr., McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-001
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Bariatric surgery; Obesity; Laparoscopic gastric bypass; Laparoscopic adjustable gastric banding
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

ARMS (3):
- Intensive Medical Management (Placebo Comparator): Medical management of obesity including medication optimization and lifestyle and dietary advice.
  Interventions: Procedure: Intensive Medical Management
- Laparoscopic Gastric Bypass (Active Comparator)
  Interventions: Procedure: laparoscopic gastric bypass surgery
- Laparoscopic Adjustable Gastric Band (Active Comparator)
  Interventions: Procedure: laparoscopic adjustable gastric banding

INTERVENTIONS:
Procedure: laparoscopic gastric bypass surgery — Laparoscopic Gastric Bypass Surgery
  Arms: Laparoscopic Gastric Bypass
Procedure: laparoscopic adjustable gastric banding — laparoscopic adjustable gastric banding
  Arms: Laparoscopic Adjustable Gastric Band
Procedure: Intensive Medical Management — lifestyle, diet, medication optimization
  Arms: Intensive Medical Management

SUMMARY:
A large number of research studies on people who were morbidly obese (extremely overweight), and had bariatric surgery (anti-obesity surgery) have shown that patients who were diabetic before surgery often experienced significant improvement in their diabetes following the surgery. For some patients, blood glucose levels returned to the normal range, and they were able to stop taking all of their diabetes medications. For others, blood glucose levels improved, allowing them to reduce their diabetes medications.

This research study is being done to determine whether bariatric surgery can safely provide better control of diabetes symptoms in obese diabetics than continuing medical management (anti-diabetic drugs in combination with diet and lifestyle changes).

There are several different types of bariatric surgery currently being used to treat morbid obesity. Two of the most common techniques are gastric bypass and adjustable gastric banding. This study will be comparing these two surgical techniques to treatment with a combination of drugs, diet, and lifestyle changes for control of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Residents of Southern Ontario, Canada
* Obese (BMI 30 to < 40 kg/m2) patients who have had type 2 diabetes mellitus for more than 5 years, complicated by at least one of the following situations that persist despite adequate management efforts. The complicating situations are:

  * Severely reduced quality of life as assessed by the Audit of Diabetes Dependent Quality of Life (ADDQoL) questionnaire
  * Metabolic lability/instability, characterized by two or more episodes of severe hypoglycemia (≤ 3mmol/L) or severe hyperglycemia (≥ 25 mmol/L), or two or more hospital visits for diabetic complications over the last year
* Despite efforts at optimal glucose control, progressive secondary complications of diabetes as defined by:

  * Retinopathy - a minimum of a three step progression using the Early Treatment Diabetic Retinopathy Study (ETDRS) grading system, or an equivalent progression as certified by an ophthalmologist familiar with diabetic retinopathy or
  * Nephropathy - persistent or progressive macroalbuminuria (>20 mg albumin/mmol creatinine) over at least 12 months (beginning anytime within the past two years) despite the use of an angiotensin-converting enzyme (ACE) inhibitor or angiotensin II receptor blocker (ARB) or
  * Neuropathy - persistent or progressing autonomic neuropathy (gastroparesis, postural hypotension, neuropathic bowel or bladder) or persistent or progressing severe peripheral painful neuropathy not responding to usual management (e.g., tricyclics, gabapentin, or carbamazepine)

Exclusion Criteria:

* Less than 18 years of age or greater than 65 years of age
* Unable to complete self and interviewer administered questionnaires in English
* Incapable of providing informed consent
* Any of the following medical conditions that may be associated with DM:

  * Recent positive history of myocardial infarction or coronary artery bypass graft or percutaneous transluminal angioplasty (less than 6 months)
  * Unstable angina pectoris
  * Recent clinically important ST-T changes on electrocardiogram (ECG) over the past year
  * Cardiac heart failure (New York Heart Association class III and IV; ejection fraction < 50%)
  * Frequent and persistent and unstable supra and ventricular arrhythmias,
  * Brain stroke, transient ischemic attack (TIA),
  * Major diabetic foot infections
  * Autonomic neuropathy resulting in orthostatic dysregulation
* History of any psychiatric illness that would make the patient a poor candidate for bariatric surgery, as determined by the study psychiatrist
* If female, pregnant or planning to become pregnant within next year
* Clinically important cancer history (impact on either lifespan or performance of lap. bariatric surgery)
* Clinically important abdominal or thoracic surgery that would impact the performance of laparoscopic bariatric procedure
* Insulin dependence for more than 10 years
* American Society of Anesthesiologists' classification of 4 or higher
* Severe gastrointestinal reflux disease with Grade 3 or 4 esophagitis
* History of pulmonary embolism or deep vein thrombosis
* Presently taking either high-dose steroids or anticoagulants
* Advanced nephropathy (Stage 4 or 5 - eGFR less than 30 ml/min)
* Any other condition that, in the opinion of the study surgeons, would make the patient a poor candidate for bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Diabetic control as assessed by HbA1c | 1 year

SECONDARY OUTCOMES:
Resolution of diabetes | 1 year
Improvement in diabetic control and cardio-metabolic profile | 1 year
Weight loss and decrease in BMI | 1 year
Reduction in the usage of insulin or other diabetic drugs | 1 year
Improvement in diabetic complications and end-organ damage | 1 year
Improvement in health-related quality of life and depression scores | 1 year
Utilization of resources and productivity losses | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Anvari, MB BS, PhD, Principal Investigator — Centre for Minimal Access Surgery, McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada